CLINICAL TRIAL: NCT04888559
Title: Effects of a Whole Grain Cereal Product on Blood Glucose Response After 3 Consecutive Meals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aventure AB (Industry)
Collaborators: Glucanova AB (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: TSP2101
Record Dates: First submitted 2021-05-04; First posted 2021-05-17 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Blood Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole grain breakfast product (Active Comparator)
  Interventions: Other: Breakfast product: Whole grain
- Reference (Placebo Comparator)
  Interventions: Other: Breakfast product: Reference

INTERVENTIONS:
Other: Breakfast product: Whole grain — This intervention is a whole grain-based breakfast product containing oats and barley.
  Arms: Whole grain breakfast product
Other: Breakfast product: Reference — This intervention is a rice-based breakfast product.
  Arms: Reference

SUMMARY:
In this pilot study it will be investigated if a whole grain product will improve the glucose response not only when it is eaten at breakfast, but also at the two following meals; lunch and dinner (2nd and 3rd meal effect) in a healthy population.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, 35 to 65 years of age
2. BMI 22-29 (±0.5) kg/m2
3. Agree to maintain consistent dietary habits and physical activity levels for the duration of the study.
4. Healthy as determined by medical history and information provided by the volunteer.
5. Willingness to complete questionnaires and follow instructions associated with the study and to complete all visits.
6. Has given voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

1. Elevated fasting blood glucose (above 6.1 mmol/L at fasting on visit 1 or 2)
2. Women who are pregnant or breast feeding
3. Any medical condition(s) or medication(s) known to significantly affect glucose metabolism. Significance to be assessed by the QI
4. Use of medication, over-the-counter medication, natural health products or dietary supplements/probiotics that may affect glucose metabolism is prohibited during this study. Significance to be assessed by the QI. Participants who are taking allowed prescribed medications must agree to maintain their current method and dosing regimen during the course of the study unless other is recommended by their physician.
5. Known Type I or Type II diabetes, including women who previously have had gestational diabetes.
6. Use of antibiotics within 2 weeks of enrollment
7. Metabolic diseases and/or chronic gastrointestinal diseases (IBS, Crohns etc.)
8. Allergy to ingredients included in investigational product, placebo, or standardized meal
9. Participants restricted to a vegetarian or vegan diet
10. Intolerance to gluten
11. Individuals who are averse to capillary blood sampling
12. Currently active smokers (or using other tobacco products, and e-cigarettes)
13. Unstable medical conditions as determined by QI
14. Participation in other clinical research trials
15. Individuals who are cognitively impaired and/or who are unable to give informed consent
16. Acute infection
17. Any other condition which in the QI's opinion may adversely affect the individual's ability to complete the study or its measures or which may pose significant risk to the individual

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
The difference in capillary blood glucose between whole grain product and reference in the total incremental area under the curve iAUC(0-120 min) for all three meals (Breakfast iAUC0-120 min + Lunch iAUC0-120 min.+ Dinner iAUC0-120 min). | Outcome measures will be assessed just before and immediately after the intervention (glucose measurements at 0-180 min after breakfast (intervention products), 0-180 min after lunch (standardized meal) and 0-120 min after dinner (standardized meal))

SECONDARY OUTCOMES:
The difference in capillary blood glucose between whole grain product and reference in the 1, 2 and 3-hour incremental area under the curve (iAUC0-60 min, iAUC0-120 min and iAUC0-180 min) after the breakfast meal. | Outcome measures will be assessed just before and immediately after the intervention (glucose measurements at 0-180 min after breakfast (intervention products)
The difference in capillary blood glucose between whole grain product and reference in the 1, 2 and 3-hour incremental area under the curve (iAUC0-60 min, iAUC0-120 min and iAUC0-180 min) after the lunch meal. | Outcome measures will be assessed just before and immediately after the intervention (glucose measurements at 0-180 min after breakfast (intervention products) and 0-180 min after lunch (standardized meal))
The difference in capillary blood glucose between whole grain product and reference in the 1 and 2-hour incremental area under the curve (iAUC0-60 min and iAUC0-120 min) after the dinner meal. | Outcome measures will be assessed just before and immediately after the intervention (glucose measurements at 0-180 min after breakfast (intervention products), 0-180 min after lunch (standardized meal) and 0-120 min after dinner (standardized meal))
The difference in capillary blood glucose between whole grain product and reference in 2-hour Cmax(0-120 min) (maximum concentration) after the breakfast, lunch and dinner meals respectively. | Outcome measures will be assessed just before and immediately after the intervention (glucose measurements at 0-180 min after breakfast (intervention products), 0-180 min after lunch (standardized meal) and 0-120 min after dinner (standardized meal))
The difference in capillary blood glucose between whole grain product and reference in 2-hour Tmax(0-120 min) (the time to maximum concentration) after the breakfast, lunch and dinner meals respectively. | Outcome measures will be assessed just before and immediately after the intervention (glucose measurements at 0-180 min after breakfast (intervention products), 0-180 min after lunch (standardized meal) and 0-120 min after dinner (standardized meal))

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Andersson, PhD, Principal Investigator — Aventure AB
Locations (1):
- Aventure AB, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No